CLINICAL TRIAL: NCT05368415
Title: Comparison Between Different Norepinephrine Bolus Doses for Management of Post-spinal Hypotension During Ceaserian Section for Patients With Preeclampsia
Brief Title: Comparison Between Three Norepinephrine Bolus Doses for Management of Post-spinal Hypotension During Ceaserian Section for Patients With Preeclampsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Arafa, lecturer of anesthesia and surgical ICU, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Levo bolus in CS
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia; Adverse Effect; Cesarean Section Complications
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 3 mcg grup (Active Comparator): this group will receive Norepinephrine bolus of 3 mcg for management of hypotension.
  Interventions: Drug: Norepinephrine
- 4 mcg group (Active Comparator): this group will receive Norepinephrine bolus of 4 mcg for management of hypotension
  Interventions: Drug: Norepinephrine
- 5 mcg group (Active Comparator): this group will receive Norepinephrine bolus of 5 mcg for management of hypotension
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — mothers will received NE bolus of 3,4 or 5 mcg for management of hypotension according to group allocation
  Other Names: levophed

SUMMARY:
Maternal hypotension after subarachnoid block is a frequent and deleterious complication during lower segment caesarean section (LSCS). Prophylaxis against hypotension using vasopressors had become a standard recommendation. In mothers with preeclampsia, post-spinal hypotension is less frequent compared to healthy mothers; thus, the latest guidelines do not recommend using vasopressors in preeclampsia patients unless there is a hypotensive episode . The incidence of post-spinal hypotension in mother with preeclampsia is nearly 25%. The commonly used vasopressors during CS are ephedrine, phenylephrine, and recently norepinephrine. The use of ephedrine is usually accompanied with maternal tachycardia and foetal acidosis. Phenylephrine (PE) had been the first line for prevention and management of maternal hypotension; however, its use in mothers with preeclampsia had not been adequately investigated. Thus, the best vasopressor for management of hypotension in mothers with preeclampsia is unknown. Norepinephrine (NE) is an alpha adrenergic agonist with weak beta adrenergic agonistic activity; thus, it does not cause significant cardiac depression as phenylephrine does. NE was introduced for use during CS with promising results when used as infusion and as boluses in healthy mothers .

The use of NE boluses in management of hypotension in preeclamptic mothers was not adequately investigated. A dose 4 mcg NE was recently evaluated in preeclamptic mothers. In this study, we will compare 3 NE bolus doses (3 mcg, 4 mcg, and 5 mcg) in management of maternal hypotension after spinal block during CS in preeclamptic mothers.

ELIGIBILITY:
Inclusion Criteria:

* pregnant female with preeclampsia
* age 18-40

Exclusion Criteria:

* age less than 18
* age above 40
* patient refusal of spinal anesthesia
* patient with eclampsia
* patient allergy to anesthesia drugs or to NE

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Neonatal concentration of HCO3 from a sample of umbilical cord as a surrogate of neonatal outcome | up to 5 minutes after delivery
  measuring HCO3 from umbilical cord blood gases analysis

SECONDARY OUTCOMES:
Rate of successful management of maternal hypotension | 2 minutes after NE bolus
  defined as returned of SBP to be > 80% of the baseline reading in the next reading 2 minutes after administration of NE bolus

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Arafa, MD, Principal Investigator — Lecturer of anesthesia and surgical ICU
Locations (1):
- Cairo university, Kasr Alainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: August 2022

REFERENCES:
- [Background] Hassabelnaby YS, Hasanin AM, Adly N, Mostafa MMA, Refaat S, Fouad E, Elsonbaty M, Hussein HA, Mahmoud M, Abdelwahab YM, Elsakka A, Amin SM. Comparison of two Norepinephrine rescue bolus for Management of Post-spinal Hypotension during Cesarean Delivery: a randomized controlled trial. BMC Anesthesiol. 2020 Apr 17;20(1):84. doi: 10.1186/s12871-020-01004-y. PMID 32303180
- [Background] Hasanin A, Amin S, Refaat S, Habib S, Zayed M, Abdelwahab Y, Elsayad M, Mostafa M, Raafat H, Elshall A, Fatah SAE. Norepinephrine versus phenylephrine infusion for prophylaxis against post-spinal anaesthesia hypotension during elective caesarean delivery: A randomised controlled trial. Anaesth Crit Care Pain Med. 2019 Dec;38(6):601-607. doi: 10.1016/j.accpm.2019.03.005. Epub 2019 Mar 30. PMID 30935897